CLINICAL TRIAL: NCT06384612
Title: The Effect Of The Use Of Pocket Cards In An Undergraduate Nursıng Course On Students' Self-Effıcacy Perceptıon And Academıc Course Success
Brief Title: The Effect Of The Use Of Pocket Cards In An Undergraduate Nursıng
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Bircan Kahraman Berberoglu, research asistant, Aydin Adnan Menderes University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Adnan Menderes U
Record Dates: First submitted 2024-04-19; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Student; Self Efficacy

STUDY DESIGN:
Intervention Model Description: experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): The control group consisted of students enrolled in the Care of a Child with Special Needs course in the 2021-2022 fall semester and enrolled in one of the branches. Students were informed about the research in the first week of the 2021-2022 fall semester, their written consent was obtained, and they were allowed to fill out the introductory information form and the Self-Efficacy Perception Scale (pre-test) in the second week. Routine course content was followed with these students throughout the course period. No intervention was made to the students. The course process was not disrupted during the research. Midterm and final exams were held on the dates determined by the faculty in order to evaluate the success of the course. The grade point averages of the students were evaluated by taking the exam table from the student information system. In the last week of the 2021-2022 fall semester, students were allowed to fill out the Self-Efficacy Perception Scale (posttest) again.
- pocket cards group (Experimental): The study group consisted of students enrolled in the Care of a Child with Special Needs course in the 2021-2022 spring semester. Introductory information form and Self-Efficacy Perception Scale were filled out. A common day was determined with the students and a 15-minute training was given on the example of preparing a pocket card. A total of nine groups of seven people were formed and they were prepared for the next week. At the end of each lesson, student groups were asked to prepare a pocket card on a 22 cm piece of paper. A WhatsApp group and an Instagram page were established to check whether the students had made their pocket cards and, if so, whether it was accurate. The cards were shared in their final form on Instagram and each student was told to turn on page notifications and like the post when they saw it so that they could instantly follow the post. In the last week, students were asked to fill out the Self-Efficacy Perception Scale again.
  Interventions: Behavioral: use of pocket cards

INTERVENTIONS:
Behavioral: use of pocket cards — Use of pocket cards of 22 cm x 11 cm size prepared by students every week in classes
  Arms: pocket cards group

SUMMARY:
The aim of this study is to examine the effect of the use of pocket cards by students taking the "Care of a Child with Special Needs" course on students' self-efficacy perceptions and course success.

1. H01. There is no difference between the self-efficacy perception scores of the students in the group who use pocket cards in the care of children with special needs course and the students in the group who do not use pocket cards.
2. H02. There is no significant difference between the course success scores of the students in the group who use pocket cards in the care of children with special needs course and the students in the group who do not use pocket cards.

DETAILED DESCRIPTION:
The research will include the parents of 194 children with special needs between the ages of 6-18, who came to four special education and rehabilitation centers in Efeler district of Aydın province between 13 September 2021 - 22 May 2022 (8 months) and were selected by stratified random sampling method.

Study data will be collected from the parents of children coming to Rehabilitation Centers and routine training by face-to-face interview technique using the child and parent information form and the Oral and Dental Health Information Evaluation Form. Data collection is expected to take approximately 15-20 minutes.

Approval will be obtained from Aydın Adnan Menderes University Faculty of Nursing Non-Interventional Research Ethics Committee to conduct the research. Permission will be obtained from the institutions to conduct the research in the centers. An explanation about the research will be made to the parents (mother or father) of the children who meet the sampling criteria, and written consent will be obtained from the parents of the children who agree to participate in the research.

While calculating the sample size, the self-efficacy perception score averages in the study titled "The effect of learning objects on academic success, self-efficacy perception, motivation and learning permanence in mathematics teaching" were used according to effect power calculation blended standard deviation. was placed on the formula and the potency was calculated (d: 13.11). Two independent groups and t test options were selected through G power analysis and power analysis was calculated according to the two-way hypothesis method. According to the previous study, when the significance level between the study group and the control group was taken as α = 0.05 and the power of the test was 1-β = 0.95, the sample size to be selected was determined as 56 people for each group. It was determined that the sample loss (students registered for the 2018-2019 spring semester who failed due to absence and failure) was approximately 15% due to the fact that among our exclusion criteria for the study were students who failed due to absence and failure. By increasing the minimum number of students planned to be included in the research and required to be in each group (n=56+0.15) by 15% (approximately 8 students), the number of samples for both groups became 64 (study group; n=64; control group n=64). It was calculated as a total of 128 students. A post-hoc power analysis will be conducted after the study. The data of the research will be analyzed using SPSS 25 (Statistical Package for the Social Sciences) program. Descriptive statistics, Chi-square test, Student-T test will be used to evaluate the study data. Student's T Test will be used to compare paired groups in the analysis of normally distributed dependent variables. Mann-Whitney U test will be applied to compare two independent data that do not show normal distribution. Values at P<0.05 will be considered statistically significant. Regression analysis will be performed to determine factors that may be related to dependent variables.

ELIGIBILITY:
Inclusion Criteria:

Taking a course on caring for a child with special needs

Exclusion Criteria:

Not preparing pocket cards for 2 consecutive weeks

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
Self-Efficacy Perception Scale | 8 months
  In order to collect data about students' self-efficacy perceptions, the 8-item self-efficacy perception scale in the motivational beliefs dimension of the "Motivational Strategies for Learning Scale" was applied. The scale is prepared as a 7-point Likert type, and the lowest score can be 8 and the highest score can be 56. Cronbach's alpha value for the Turkish form of the self-efficacy perception scale was found to be 0.92. In order to use the Self-Efficacy Perception Scale, permission will be requested via e-mail from author, who carries out the validity and reliability of the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Hüsniye çalışır, PHD, Study Chair — Aydın Adnan Menderes Univercity
Locations (1):
- Bircan Kahraman Berberoğlu, Efeler, Aydın, Turkey (Türkiye)